CLINICAL TRIAL: NCT02797639
Title: The Effectiveness of Collaborative Consultation for Participation Among Students With Moderate Intellectual Disability (Co-PID)
Brief Title: Collaborative Consultation for Participation Among Students With IDD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ono Academic College (Other)
Responsible Party: Principal Investigator, Efrat Selanikyo, Lecturer, Ono Academic College
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: Onoac
Record Dates: First submitted 2016-05-28; First posted 2016-06-13 (Estimated); Last update posted 2016-06-14 (Estimated); Status verified 2016-06

CONDITIONS: Mental Retardation and Developmental Disabilities With Organic Condition
Keywords: Intellectual Disability; Collaborative Consultation; Participation
MeSH Terms: conditions — Intellectual Disability

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Co-PID (Experimental): Eight collaborative consultation meetings between occupational therapist to each teacher in purpose of enhancing participation of students in class
  Interventions: Other: Co-PID
- In-service (Active Comparator): Three in- service meetings to all homeroom teachers together, in purpose of enhancing participation of students in class
  Interventions: Other: IS

INTERVENTIONS:
Other: Co-PID — The program was carried out by the school occupational therapist and homeroom teachers. The Co-PID had two phases. The first phase was a 1.5 hour in-service meeting that focused on the concept of "Participation".
  In the second phase of the Co-PID intervention, a collaborative consultation model was used. It included eight 45-minute consultation meetings, which took place every other week over a 3-months period. The meetings took place between the occupational therapist and each teacher, with the purpose of brainstorming; thinking of activities that the teacher could implement during the lessons for enhancing participation among the students.
  Arms: Co-PID
Other: IS — IS group included three meetings, a 1.5 hour in-service meeting focusing on the concept of participation, and two more workshop meetings aimed at sharing teachers' experience.
  Arms: In-service

SUMMARY:
Objective: Developing and corroborating the Collaborative Consultation for Participation of Students with Intellectual Disability (Co-PID) program, for enhancing classroom participation among students with moderate Intellectual and Developmental Disability (IDD).

Method: study took place in two special education schools and included students with moderate IDD (n=60) and their teachers (n=11). The settings were randomly assigned to intervention or control group. In the intervention group, Co-PID program was employed; in the control group an In-Service (IS) was employed. Participation was evaluated at pre-test and post-test.

DETAILED DESCRIPTION:
The study was conducted in three phases: (a) pre-test; (b) intervention; and (c) post-test

Pre-test. Using the 'Structured Observation of Students' Participation in Class', each student in both groups was observed four times during different lessons (with a 1-week interval between observations) to establish a baseline for level of participation. All pre-test observations were conducted between the 2nd and 3rd months of the school year, by an occupational therapist with 8 years of experience working with children with developmental delays. The observer was trained in using the 'Structured Observation of Students' Participation in Class' and was not blinded to the schools' assignment (Co-PID or IS). During this period the teachers, who were blinded to the school assignment, were asked to teach in a regular manner without changing the content or design of their lessons. Next, the teachers filled out the School Function Assessment questionnaire for each student. Finally, based on the 'Structured Observation of Students' Participation in Class' scores and teachers' familiarity with the students' function, the occupational therapist and each of the participating teachers jointly filled-out the 'Goal Attainment Scaling' form. Each student had three goals, one for each of the participation skills: Communicating, Choosing and Initiating. Post-test. This phase was conducted during the 9th and 10th months of the school year, and was identical to the pre-testing phase in terms of both process and measures used

ELIGIBILITY:
Inclusion Criteria:

1. A diagnosis of moderate IDD
2. Mobility independence
3. No secondary diagnosis of autism, nor sensory disabilities such as blindness or deafness
4. Students had been studying at the school for at least one year prior to data collection.

Exclusion Criteria:

-

Ages: 7 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2014-09; Primary Completion 2015-08 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Structured Observation of Students' Participation in Class | within one month after intervention completion
  A structured observation for examining participation of students with moderate IDD in the classroom. It includes 25 items that focus on three classroom participation skills: (a) Communicating (listening and expressing; 7 statements); (b) Choosing (8 statements), and (c) Initiating (10 statements). The observer rates the active participation of students during an entire lesson (about 45 minutes), with regards to each of the items, on a scale of 0 (Does not participate) to 4 (Fully participates). In addition, each statement includes a 'Not relevant' option - when the student was not given the opportunity to perform the task.

SECONDARY OUTCOMES:
School Function Assessment Questionnaire "through study completion" | within one month after intervention completion
  a criterion-referenced, standardized assessment that measures students' performance in functional tasks that support their participation in the school program. The School Function Assessment includes three parts: (a) Participation, (b) Task supports and (c) Activity performance. It is completed by one or more school professionals who are highly familiar with the students being observed.
Goal Attainment Scaling "through study completion" | within one month after intervention completion
  a method for scoring the extent to which the client's goals are achieved in the course of intervention. Functional goals are determined through a collaborative process between clinician and client or caregiver, prior to intervention. Scoring is based on a scale, where the user breaks-down each goal's performance on a 5-point scale ranging from -2 to 2

CONTACTS AND LOCATIONS:
Overall Officials: Naomi Weintraub, Prof, Study Director — Hebrew University

IPD SHARING:
Plan to Share IPD: No